CLINICAL TRIAL: NCT03569189
Title: Impact of Short-term Overfeeding With a Saturated Fat-rich Diet on Fasted Systemic and White Adipose Tissue Inflammatory Responses
Brief Title: Impact of a High Saturated Fat Diet on Fasted Systemic and White Adipose Tissue Inflammatory Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Oonagh Markey, Principal Investigator, Loughborough University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R18-P040
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Inflammation; Obesity; Inflammatory Response; Cardiovascular Diseases
MeSH Terms: conditions — Inflammation; Obesity; Cardiovascular Diseases | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Fat Diet (Experimental): Participants will consume a high-fat, high-calorie diet for 7 days (i.e. westernised diet) following a 3-day weight maintenance diet. Measurements will be made pre- and post-high fat diet intervention.
  Interventions: Other: High Fat Diet

INTERVENTIONS:
Other: High Fat Diet — Participants will consume a high fat diet for 7 days with 65% of energy from fat. The diet will also provide an energy excess at 150% of energy requirements.
  Participants will be provided with all of their meals and snacks throughout the study.

SUMMARY:
This study will investigate the effect of a 7-day westernised high-fat (65% of kilocalories), high-calorie (150% of requirements) diet on markers of inflammation in the blood and white adipose tissue. Participants will firstly complete a 3-day weight maintenance phase (Days 1-3) before completing a 7-day high fat diet intervention (Days 4-10). On days 4 and 11 participants will complete a laboratory visit where anthropometric measurements, blood and adipose samples will be collected.

The investigators hypothesise that consuming a high-fat, high-calorie diet for 7 days will alter the inflammatory responses in white adipose tissue and will induce metabolic endotoxaemia / systemic inflammation.

ELIGIBILITY:
Inclusion criteria:

* 18-40 years
* BMI = 21.0-29.9 kg/m2
* Male or female
* Physically active (> 3 x 30 min moderate exercise per week)
* Healthy
* No cardiometabolic (e.g. heart disease, high blood pressure, type 2 diabetes) or inflammatory illness

Exclusion criteria:

* Inactive (< 3 x 30 min moderate exercise per week)
* Smoker
* Women who are pregnant or lactating
* Medication/supplements known to interfere with study outcomes or prescribed antibiotics within the last 3 months
* Unstable weight history (≥3kg loss or gain in the previous 3 months)
* An allergy to lidocaine
* Food allergies (e.g. gluten, dairy) and intolerances (e.g. lactose) which could impede compliance to the diet
* Vegetarian/ vegan (as the high-fat diet is based on animal fats)
* Consumption of probiotics yogurts during or within the four weeks prior to the start of the study (e.g. Actimel, Activia, Yakult, Yeo Valley)
* Alcohol consumption >28 units per week for a man (i.e. not more than 14 pints of beer or 28 small glasses of wine) or >21 units per week for a woman (i.e. more than 10 and a half pints of beer or 21 small glasses of wine)
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention or metabolic study
* Restrained eaters (determined by Three Factor Eating Questionnaire)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Protein expression (content and phosphorylation) of key markers of metabolic inflammation in white adipose tissue (for example assessment of NFKB/IKBa total protein and phosphorylation by western blot analysis) | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  This will be assessed following the collection of fasted white adipose tissue samples

SECONDARY OUTCOMES:
Systemic Markers of Inflammation (for example CRP, TNFa and IL-6 concentrations, determined by spectrophotometric assay/ ELISA) | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  Assessed following the collection of fasted blood samples
Gene expression of key markers of metabolic inflammation in white adipose tissue | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  This will be assessed following the collection of fasted white adipose tissue samples
Fasting Serum Markers of Insulin Resistance (for example insulin and glucose concentrations, determined using an ELISA/ spectrophotometric assay) | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  Assessed following the collection of fasted blood samples
Fasting Serum Lipid Profile (for example total, HDL and LDL cholesterol, TAG and NEFA concentrations, measured using a spectrophotometric assay) | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  Assessed following the collection of fasted blood samples
Systemic Markers of Metabolic Endotoxemia (for example LBP and sCD14 concentrations, determined using an ELISA) | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  Assessed following the collection of fasted blood samples
Immune Cell Populations in the Blood | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  Assessed following the collection of fasted blood samples
Anthropometric Measurements (for example height and weight that will be aggregated to report BMI in kg/m^2) | Change between pre- and post-high fat diet (assessed on days 4 and 11)
  Measured using standard equipment
Physical Activity | Habitual physical activity will be assessed for 3 days prior to commencing the high-fat diet intervention (days 1-3) and during the final 3 days of the intervention (days 8-10)
  Assessed using Actigraph accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Oonagh Markey, BSc, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Dewhurst-Trigg R, Wadley AJ, Woods RM, Sherar LB, Bishop NC, Hulston CJ, Markey O. Short-term High-fat Overfeeding Does Not Induce NF-kappaB Inflammatory Signaling in Subcutaneous White Adipose Tissue. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa158. doi: 10.1210/clinem/dgaa158. PMID 32232380